CLINICAL TRIAL: NCT02693613
Title: Pharmacokinetic Study of ASP1517 - Evaluation of the Effect of Kremezin® on the Pharmacokinetics of ASP1517 in Non-elderly Healthy Adult Male Subjects, When Administered Concomitantly or in a Time Separated Manner.
Brief Title: Pharmacokinetic Study of ASP1517 With Kremezin®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0204
Record Dates: First submitted 2016-02-03; First posted 2016-02-29 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
Keywords: Drug-drug interaction; Kremezin; Pharmacokinetics; ASP1517
MeSH Terms: interventions — AST 120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Treatment arm includes 4 periods, single dose of ASP1517 alone, single dose of ASP1517 + Kremezin® without a time lag, single dose of ASP1517 + Kremezin® with a time lag (1 h before ASP1517 administration) and single dose of ASP1517 + Kremezin® with a time lag (1 h after ASP1517 administration)
  Interventions: Drug: ASP1517; Drug: Kremezin®
- Group 2 (Experimental): Treatment arm includes 3 periods, single dose of ASP1517 alone, single dose of ASP1517 + Kremezin® with a time lag (2 h before ASP1517 administration) and single dose of ASP1517 + Kremezin® with a time lag (2 h after ASP1517 administration)
  Interventions: Drug: ASP1517; Drug: Kremezin®

INTERVENTIONS:
Drug: ASP1517 — Oral
Drug: Kremezin® — Oral

SUMMARY:
The objective of this study is to evaluate the effect of Kremezin® on the pharmacokinetics of single dose of ASP1517 in healthy non-elderly adult male subjects when administered concomitantly or in a time separated manner.

ELIGIBILITY:
Inclusion Criteria:

* Body weight (at screening): ≥50.0 kg and <80.0 kg
* Body-mass index (BMI) (at screening): ≥17.6 and <26.4 kg/m2
* Subject must agree to use contraception consisting of two established forms (1 of which must be a barrier method) starting at the time of informed consent and continuing throughout the treatment period and for 84days after ASP1517 administration in the last period:
* Subject must agree not to donate sperm starting at the time of informed consent and continuing throughout 84 days after the last administration of ASP1517 in the last period.

Exclusion Criteria:

* Received or is scheduled to receive any investigational drugs in other clinical trials or post-marketing studies within 120 days before screening or during the period from screening to the hospital admission day of the Period 1 (Day -1).
* Received or is scheduled to receive medications (including over-the-counter [OTC] drugs) within 7 days before the hospital admission day of the Period 1 (Day -1).
* Received or is scheduled to receive supplements within 7 days before the hospital admission day of the Period 1 (Day -1).
* Deviates from any of the normal range of blood pressure, pulse rate, body temperature and standard 12-lead electrocardiogram (ECG) specified at screening or the hospital admission day of the Period 1 (Day -1).
* Meets any of the following criteria for laboratory tests at screening or the hospital admission day of the Period 1 (Day -1). Normal ranges of each test specified at the study site or the test/assay organization will be used as the normal ranges in this study.
* Concurrent or previous drug allergies.
* Development of (an) upper gastrointestinal symptoms within seven days before the hospital admission day of the Period 1 (Day -1).
* Concurrent or previous hepatic disease, heart disease, respiratory disease, gastrointestinal disease, gastrointestinal obstruction,oesophageal varices, renal disease, endocrine disease, cerebrovascular disorder, malignant tumor, retinal neovascular lesions and macular edema.
* Concurrent chronic constipation or diarrhoea.
* A history of digestive tract excision.
* Previous use of hypoxia inducible factor-prolyl hydroxylase inhibitors (HIF-PHI) such as ASP1517 (FG-4592), YM311 (FG-2216) or erythropoietin products.
* Excessive alcohol or smoking habit.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of ASP1517: AUCinf | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameter of ASP1517: Cmax | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  Cmax: Maximum concentration

SECONDARY OUTCOMES:
PK parameters of ASP1517: AUClast | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  AUClast: Area under the concentration-time curve from the time of dosing extrapolated to the last measurable concentration
PK parameters of ASP1517: CL/F | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  CL/F: Apparent total systemic clearance
PK parameters of ASP1517: t1/2 | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  t1/2: Terminal elimination half-life
PK parameters of ASP1517: tmax | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  tmax: Time of Cmax
PK parameters of ASP1517: tlag | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  tlag: Time point prior to the time point corresponding to the first measurable (non-zero) concentration
PK parameters of ASP1517: Vz/F | Pre-dose, 0.5, 1, 2, 3, 5, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hr after dosing
  Vz/F: Apparent volume of distribution during the terminal elimination phase
Safety assessed by Adverse events | Up to 72 hours after final study drug dosing
Safety assessed by Vital signs | Up to 72 hours after each study drug dosing
  Supine blood pressure, supine pulse rate and axillary body temperature
Safety assessed by Laboratory tests | Up to 72 hours after each study drug dosing
  Hematology, blood biochemistry and urinalysis
Safety assessed by Standard 12-lead ECG | Up to 72 hours after each study drug dosing
  ECG: Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided